CLINICAL TRIAL: NCT05718791
Title: CXC-chemokine Ligand 9 (CXCL9) and Endothelial Activation and Stress Index (EASIX) for Prediction of Acute Graft Versus Host Disease
Brief Title: CXCL9 and EASIX for Prediction of Acute Graft Versus Host Disease
Status: Recruiting | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Shatha Farhan, Clinical Assistant Professor, Henry Ford Health System
Other Study IDs: hhf
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: GVHD,Acute
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood sample — blood sample to check CXCL9 and EASIX at day 28 post stem cell transplant

SUMMARY:
The prediction of severe acute GVHD before it occurs is of high importance for ensuing clinical decisions and overall success of allogeneic SCT. The key immunologic signatures associated with clinical outcomes after different graft versus host disease prophylaxis methods or peripheral blood stem cell transplant are largely unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 year old admitted for allo SCT PB for malignant disease.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients >18 year old admitted for allo SCT PB for malignant disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
predictors of acute GVHD | CXCL9 combined with EASIX calculated at day 28 +/- 2 post SCT can be used as predictors of acute GVHD by day 100.
  CXCL9 combined with EASIX can be used as predictors of acute GVHD

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States